CLINICAL TRIAL: NCT02261038
Title: Comparative Study pf the Femoral Prothesis-rotation in Conventional X-Ray, in Axial CT Slices and 3D-reconstructed CT
Brief Title: Comparison of the Femoral Prothesis-rotation in Conventional X-ray, in Axial CT Slices and 3D-reconstructed CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Tobias Hirschmann (Other)
Responsible Party: Sponsor-Investigator, Michael Tobias Hirschmann, PD Dr. med., Kantonsspital Baselland Bruderholz
Organization: Kantonsspital Baselland Bruderholz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rad-2CT-3CT_001_MH; 332/13 (Other: Ethikkommission Nordwest- und Zentralschweiz)
Record Dates: First submitted 2014-07-28; First posted 2014-10-10 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; total knee prothesis; X-Ray; Kanekasu radiographs; femoral component rotation; effects
MeSH Terms: conditions — Osteoarthritis | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kanekasu radiographs (Other): No drugs or devices are used in this study. Commonly available radiological techniques such as radiographs and CT are used. All patients undergo a CT of the knee and a special radiograph (Kanekasu technique).
  Interventions: Other: Kanekasu radiographs

INTERVENTIONS:
Other: Kanekasu radiographs — No interventions are performed here. All patients undergo CT and special radiographs of the knee to assess femoral TKA rotation.
  Other Names: Femoral component rotation; total knee prothesis; X-ray; kanekasu-technic

SUMMARY:
Femoral component rotation in total knee arthroplasty (TKA) has been considered an important factor for outcome. However, measurement of femoral component rotation is difficult to perform.

Femoral TKA component rotation can be assessed on special radiographs (Kanekasu technique), axial CT slices and 3D reconstructed CT images.

It was the hypothesis that measurements on radiographs are comparable to measurement on CT images.

Measurements of femoral TKA rotation will be measured three times by three different observers and inter- and intraobserver reliability is calculated. The absolute values of each measurement method is noted in degrees.

DETAILED DESCRIPTION:
Femoral component rotation in total knee arthroplasty (TKA) has been considered an important factor for outcome. However, measurement of femoral component rotation is difficult to perform.

Femoral TKA component rotation can be assessed on special radiographs (Kanekasu technique), axial CT slices and 3D reconstructed CT images.

It was the hypothesis that measurements on radiographs are comparable to measurement on CT images.

In agreement with our standard diagnostic algorithm for patients with pain and problems after TKA CT images as well as Kanekasu radiographs are performed. If the Kanekasu radiograph is comparable reliable, it could be possible to use this radiograph instead.

Measurements of femoral TKA rotation will be measured three times by three different observers and inter- and intraobserver reliability is calculated. The absolute values of each measurement method is noted in degrees. The measurements are performed with two weeks interval and the different observers are blinded to their previous and the measurements of the others.

The absolute difference of femoral TKA rotation is calculated between and inter the groups investigated.

Intra class correlation coefficients are calculated for inter- and intraobserver reliability.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee prosthesis (primary)
* >55 years

Exclusion Criteria:

* pregnancy
* lactating women

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Femoral TKA component rotation in degrees | one year
  Femoral TKA component rotation in degrees is assessed on radiographs (Kanekasu), axial CT and 3D reconstructed CT images. All three measurement by each three observers are compared to each other.

SECONDARY OUTCOMES:
Inter- and intraobserver reliability of TKA femoral component rotation | one year
  Inter- and intraobserver reliability of TKA femoral component rotation are calculated by intra class correlation coefficients (ICC) and compared between all three measurement methods.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Hirschmann, MD, Principal Investigator — Dept. of Orthop. Surgery and Traumatology, Kantonsspital Baselland - Bruderholz, Unitverstity of Basel, Switzerland
Locations (1):
- Kantonsspital Baselland, Bruderholz, Bruderholz, Basel-Landschaft, Switzerland